CLINICAL TRIAL: NCT01785225
Title: Ultrasound-guided Blood Sampling With a Sterile and Dry Puncture Area
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Aarhus University Hospital (Other)
Collaborators: Danish Cancer Society (Other)
Responsible Party: Principal Investigator, Sofie Thorn, Research year student, Aarhus University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 1-10-72-589-12
Record Dates: First submitted 2013-02-01; First posted 2013-02-07 (Estimated); Last update posted 2013-02-07 (Estimated); Status verified 2013-02

CONDITIONS: Ultrasound; Sterile Puncture Area; Blood Sampling

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- modified commercial drape Tegaderm (R) (Experimental)
  Interventions: Device: A product type of the modified commercial drape Tegaderm (R)

INTERVENTIONS:
Device: A product type of the modified commercial drape Tegaderm (R) — We test if a product type of the modified commercial drape Tegaderm(R) can bee used when taking blood samples under the guidance af ultrasound. The drape is used to keep the puncture area sterile and clean of ultrasound gel.
  Other Names: Drape: Tegaderm(R) Film (3M, USA).

SUMMARY:
Thousands of vein punctures are done every day at hospitals worldwide. Vein puncture are performed in connection with blood sampling, peripheral intravenous catheter (PIV) placement or blood donation. The predominantly used venous for blood withdraw are in the cubital region because in this area venous are most superficial placed and most often visible for the human eye. However, when using the usual blind landmark and palpation method in this region, it often proves exceedingly difficult or even impossible to obtain peripheral venous access on patients who are obese, chronically ill, hypovolemic or intravenous drug users. Various studies have shown that the success rate for establishing a vascular access with ultrasound compared to blind landmark technique is higher in patients with difficult access. When ultrasound is used to establish intravascular access, the prerequisite sterile puncture area can be challenging to meet due to ultrasound gel on the area and the fact that the ultrasound transducer cannot be wiped clean with alcohol after being in contact with a patient's skin or blood. A strict sterile procedure is important to reduce complications related to infection.The traditional way of coping with this is by covering the transducer and the wire in a long sterile sheet and using sterile gel. The sheet must be tight with rubber band around the transducer and pulled tightly around the transducer foot to prevent artefacts from appearing on the screen. This is an expensive and time consuming method, and it still leaves the problem with gel in the puncture area.

The investigators have developed a method by where all these problems are solved by using, a slightly modified, commercial drape in combination with the Dynamic Needle Tip Positioning technique

The investigators hypothesize that it is possible to perform ultrasound-guided venous puncture with a sterile and dry puncture area and that puncture can be performed proximal and distal to the traditional puncture side.

It is a procedure presenting study that serves to demonstrate the feasibility of the method in ten healthy volunteers. The study will take place at Aarhus University Hospital, Skejby.

ELIGIBILITY:
Inclusion Criteria:

* age between 18 and 70 years of age
* mentally competent
* of good health

Exclusion Criteria:

* age below 18 or above 70 years of age
* daily use of blood thinner medication
* suffering from a chronic illness that requires frequent blood withdrawals
* heart conditions or vascular diseases
* People known to experience vasovagal episodes when having blood samples taken

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2013-02; Primary Completion 2013-03 (Estimated); Study Completion 2013-03 (Estimated)

PRIMARY OUTCOMES:
Number of successful blood withdrawals | During blood sampling

SECONDARY OUTCOMES:
Image quality with and without sterile cover | During blood sampling

OTHER OUTCOMES:
Number of skin penetrations needed to puncture the vein | During blood sampling
Unexpected difficulties with the sterilization procedure | during blood sampling
  Does the Tegaderm (R) device provide adequate protection so no gel will get into the puncture area? Is it possible to move the probe as the operator desires despite of the Tegaderm (R) device?
Number of posterior vessel wall punctures | during blood sampling
Time spent from tourniquet is placed to blood withdrawals | during blood sampling

CONTACTS AND LOCATIONS:
Overall Officials: Erik Sloth, Professor, MD, Study Director — Aarhus University Hospital
Locations (1):
- Aarhus University Hospital, Skejby, Aarhus, Denmark